CLINICAL TRIAL: NCT01191398
Title: Effectiveness of Atropine and Glycopyrrolate to Reduce Hyper Salivation With Ketamine Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig J. Huang (Other)
Responsible Party: Sponsor-Investigator, Craig J. Huang, Associate Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 012008-058
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Results first posted 2014-03-20 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Sialorrhea
Keywords: Hypersalivation; Conscious Sedation; Procedural Sedation; Ketamine; Atropine; Glycopyrrolate
MeSH Terms: conditions — Sialorrhea | interventions — Atropine; Glycopyrrolate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo and Ketamine (Placebo Comparator): Normal Saline 0.9% will act as a placebo. Two ml of normal saline 0.9% will be administered intravenously 30 minutes prior to the administration of the ketamine.
  Interventions: Drug: Normal saline 0.9%
- Atropine and Ketamine (Active Comparator): Atropine will be administered as a single dose of 0.01 mg/kg, with a minimum of dosage of 0.1 mg and a maximum dosage of 0.4 mg, intravenously 30 minutes before the administration of the ketamine.
  Interventions: Drug: Atropine (0.01mg/kg)
- Glycopyrrolate and Ketamine (Active Comparator): Glycopyrrolate will be administered as a single dose of 0.01 mg/kg, with no minimum dosage and a maximum dose of 0.4 mg, intravenously 30 minutes before the administration of the ketamine.
  Interventions: Drug: Glycopyrrolate (0.01mg/kg)

INTERVENTIONS:
Drug: Atropine (0.01mg/kg) — Atropine will be given at 0.01mg/kg with a minimum dosage of 0.1mg and a maximum dosage of 0.4mg. This medication will be given once by IV 30 minutes before the administration of Ketamine.
  Other Names: AtroPen; Atropine sulfate
  Arms: Atropine and Ketamine
Drug: Glycopyrrolate (0.01mg/kg) — Glycopyrrolate will be given at 0.01mg/kg with no minimum dosage and a maximum dosage of 0.4mg. This medication will be given once by IV 30 minutes before the administration of Ketamine.
  Other Names: Robinul
  Arms: Glycopyrrolate and Ketamine
Drug: Normal saline 0.9% — Normal Saline of 0.9% will be given at a volume of 2mL. This medication will be given once by IV 30 minutes before the administration of Ketamine
  Other Names: 0.9% Sodium Chloride
  Arms: Placebo and Ketamine

SUMMARY:
The purpose of this study is to determine if the antisialagogues (anti-salivary agents), Atropine and Glycopyrrolate, are effective in reducing hypersalivation when sedating patients with Ketamine for procedural sedation in the emergency department or abscess clinic. The investigators will measure salivary flow rate by collecting oral secretions by oral suctioning over a 30 minute time period starting with the administration of Ketamine. The investigators hypothesize that patients who receive either atropine or glycopyrrolate will have fewer oral secretions than patients who receive placebo.

DETAILED DESCRIPTION:
Ketamine is a common sedation agent used in the pediatric emergency department for a variety of procedures, used in clinical practice since 1970. One potential side effect of Ketamine is hypersalivation, potentially leading to laryngospasms. To prevent hypersalivation (and reduce the potential for laryngospasms), an anti-salivary agent, such as Atropine, is commonly given in combination with Ketamine. Recently, however, the necessity of this practice has been brought into question. The consideration of using a different drug, glycopyrrolate, has been debated. The purpose of this study is to compare the effectiveness of each medication in addition to the placebo control.

Patients enrolled into this study must present to the emergency department or abscess clinic with the need to receive Ketamine as part of a sedation procedure (as determined by the treating physician). This study will randomize enrolled patients to receive double-blinded Atropine, Glycopyrrolate or placebo given 30 minutes prior to Ketamine. After Ketamine is administered, a trained medical person will suction the patient's mouth every 5 minutes for a total of 30 minutes, collecting all oral secretions. Total saliva production will be measured and salivary flow rates will be calculated and compared between each assigned group. Adverse events and complications will be monitored throughout the patient's stay in the emergency department or abscess clinic.

ELIGIBILITY:
Inclusion Criteria:

* Children age 6 months to 18 years (inclusive) presenting to Children's Medical Center Emergency Department or Abscess Clinic.
* Children whom the attending physician feels need procedural sedation with the intravenous medication, Ketamine.

Exclusion Criteria:

* Children who are ASA class III or greater.
* Children with an allergy or contraindication to ketamine, atropine or glycopyrrolate.
* Inability to tolerate oral suctioning.
* Any condition or situation whereby the patient would be unable to have his/her head turned to one side.
* Patient history of vomiting or diarrhea in the last 24 hours
* Patients who have taken an anti-sialogogue within the previous 24 hours.
* Patients that need to receive Midazolam or other benzodiazepines.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2010-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Rodriguez, MD, Study Chair — University of Texas Southwestern Medical Center; Craig Huang, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children's Medical Center at Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Normal Saline0.9% will act as a placebo.
  Placebo: Normal Saline of 0.9% will be given at a volume of 2mL. This medication will be given once by IV 30 minutes before the administration of Ketamine
- Atropine: Atropine (0.01mg/kg): Atropine will be given at 0.01mg/kg with a minimum dosage of 0.1mg and a maximum dosage of 0.4mg. This medication will be given once by IV 30 minutes before the administration of Ketamine.
- Glycopyrrolate: Glycopyrrolate (0.01mg/kg): Glycopyrrolate will be given at 0.01mg/kg with no minimum dosage and a maximum dosage of 0.4mg. This medication will be given once by IV 30 minutes before the administration of Ketamine.
Period: Overall Study
Arm/Group | Placebo | Atropine | Glycopyrrolate
Started | 17 | 17 | 18
Completed | 17 | 17 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Atropine | Glycopyrrolate | Total
Number analyzed (Participants) | 17 | 17 | 18 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.34 (4.07) | 5.09 (3.76) | 4.48 (3.09) | 4.85 (3.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 11 | 25
  Male | 11 | 9 | 7 | 27
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 18 | 52

OUTCOME MEASURES:

1. Primary Outcome: Difference in Salivary Flow Rate (ml/Min) Between Study Groups
Description: Oral Secretions will be collected by oral suctioning starting at the time Ketamine is administed until 30 minutes post Ketamine administration. Suctionings will be done by trained personnel every 5 minutes starting with the Ketamine administration. Flow rate will be calculated by dividing the total volume of saliva suctioned by the total time suctioned (30 minutes)
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Placebo | Atropine | Glycopyrrolate
Number analyzed (Participants) | 17 | 17 | 18
ml/min | .072 (0.111) | .003 (0.0084) | NA (NA) — No detectable measurable amount was collected, so mean and SD could not be calculated.

2. Secondary Outcome: Monitoring of Adverse Events During Study Administration
Description: Subjects will be monitored for episodes of apnea, laryngospasm, vomiting, oxygen desaturation(<92%), and changes in heart rate and blood pressure. The time frame will include the time the study medication is administered until at least 30 minutes post Ketamine administration.
Time Frame: 1 hour
Measure: Number; unit: adverse events
Arm/Group | Placebo | Atropine | Glycopyrrolate
Number analyzed (Participants) | 17 | 17 | 18
adverse events | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Placebo | Atropine | Glycopyrrolate
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 1/17 | 0/17 | 0/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Atropine (N=17) | Glycopyrrolate (N=18)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Episode of vomiting, post sedation. However, patient able to tolerate oral intake prior to hospital discharge.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No